CLINICAL TRIAL: NCT01817712
Title: CSP #589 - Veterans Individual Placement and Support Towards Advancing Recovery
Brief Title: Veterans Individual Placement and Support Towards Advancing Recovery
Acronym: VIP-STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 589
Record Dates: First submitted 2013-03-20; First posted 2013-03-25 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Posttraumatic neuroses; posttraumatic stress disorder; PTSD; Supported employment; IPS; CWT; TWP; Individual placement and support; Compensated work therapy; Transitional work program
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Palliative Care; Employment, Supported; Myo-Inositol-1-Phosphate Synthase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual Placement and Support (IPS) (Experimental): The IPS intervention must achieve a rating of >66 of a possible 75 points on the Supported Employment Fidelity Scale. The fidelity ratings are conducted by the National IPS Fidelity Monitor at biannual on-site monitoring visits.
  Interventions: Behavioral: Individual Placement & Support
- VA Transitional Work Program (TWP) (Active Comparator): TWP will adhere to a lower rating (less than or equal to 55 of a possible 75 points) on the Supported Employment Fidelity Scale rated by the National Fidelity Monitor. The TWP specialist participates in face-to-face supervision with the local Compensated Work Therapy (CWT) team according to the CWT manager's schedule.
  Interventions: Behavioral: VA Transitional Work Program

INTERVENTIONS:
Behavioral: Individual Placement & Support — IPS uses an integrated "place-train" approach to help people obtain and maintain community-based competitive employment in their chosen occupation.
  Other Names: Supported Employment, IPS
  Arms: Individual Placement and Support (IPS)
Behavioral: VA Transitional Work Program — The long-standing approach to vocational rehabilitation in VHA and state programs is the "train-place" or "stepwise" model that is founded on the assumption that the patient or client benefits from some form of pre-vocational training, instruction, or practice in a protected, but artificial, work setting prior to entering or being placed in a competitive work role.
  Other Names: TWP
  Arms: VA Transitional Work Program (TWP)

SUMMARY:
The primary objective of CSP#589 VIP-STAR is to evaluate the effectiveness of Individual Placement & Support (IPS) in unemployed Veterans with PTSD. The primary hypothesis is that, compared to those treated with transitional work program (TWP), unemployed Veterans with PTSD treated with IPS will be significantly more likely to become a steady worker. A steady worker is defined as holding a competitive job for greater than or equal to 50% of the 18-month study follow-up period (i.e., greater than or equal to 39 of the 78 weeks). All participants will be followed for 18 months post-randomization.

12/14/12: Analytic plan augmented to allow for a sensitivity analysis of the primary outcome that would exclude the first 12 weeks post-randomization, and evaluate between group proportion of steady worker status, as defined by working in a competitive job for greater than or equal to 50% of the weeks during week 13-78.

7/1/13: Analysis plan has been augmented to include a logistic regression analysis of the primary outcome, adjusted for participating medical center.

10/4/13: Addition of the IPS-25 Fidelity Scale. The addition of the IPS-25 scale should increase the validity of study results.

1/15/15: Addition of an Interactive Voice Recognition/Web-based (IVR/Web) System; as an option for weekly data capture of the primary outcome data (employment history).

8/17/15: Approval of Supplemental Data Collection at Participant Study Exit; use of the data collected will supplement the study analysis plan and, provide further insight into the impact of vocational rehab. A Participant Satisfaction Survey will allow study participants to indicate their level of satisfaction with the study, vocational rehabilitation intervention and, suggestions for future research.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) affects more than 600,000 US Veterans and is the most common psychiatric condition for which Veterans seek VA disability benefits, making up a substantial proportion of the $23 billion pensions and disability annual budget. Although many Veterans with PTSD are college educated, few have jobs, almost 40% are impoverished, and most report work, role and social functioning scores below those of persons with serious mental illness. Veterans returning from the Gulf War-era II conflicts, defined as having served in the military since Sept 2001, often experience PTSD and confront unemployment upon their military discharge. According to a March 2011 report from the U.S. Department of Labor, the 2010 unemployment rates were 11.5% for these Gulf War-era II Veterans, 21% for service-connected disabled Gulf War-era II Veterans, 13% for all service-connected Veterans of all eras combined and 9.4% for non Veterans. The current methods used by the VA Compensated Work Therapy (CWT) programs do not sufficiently meet the employment rehabilitation needs of Veterans with PTSD. In a VA Northeast Program Evaluation Center (NEPEC) study evaluating administrative data of 5,862 Veterans from 122 CWT programs, Veterans with PTSD were 19% less likely to be employed at discharge from the VA CWT program compared to those without a diagnosis of PTSD. The rate of competitive employment at discharge was only 30% for Veterans with PTSD. Similarly, another VA study found that Veterans with PTSD involved in CWT were no more likely to be employed at 4 months follow-up compared to those who participated in a specialized PTSD treatment program.

Over the past two decades of studies, the Individual Placement and Support (IPS) model of Supported Employment has yielded remarkably robust and consistent employment outcomes for individuals with serious mental illness (defined as schizophrenia, schizoaffective disorder, bipolar disorder, and major depression with psychotic features). Overall, approximately two-thirds of participants in clinical trials with serious mental illness who received IPS achieved competitive employment. However, Veterans with PTSD have very different clinical characteristics and employment challenges compared to Veterans with SMI. Serving as the first study in a PTSD population, a recent single site pilot study found superior outcomes from IPS compared to the conventional VA vocational rehabilitation program (VRP) in unemployed Veterans with PTSD (n=85). During the 12-month study follow-up period, 76% of the Veterans with PTSD randomized to IPS gained competitive employment, compared to 28% of those randomized to VRP. Together with the evidence base accumulated in the serious mentally ill population, the positive results of the pilot study in PTSD support a VA Cooperative Study to definitively test the effectiveness of IPS in Veterans with PTSD.

As the primary outcome, the two groups will be compared in terms of the proportion of study participants who met the definition of steady worker, i.e., hold competitive employment for at least 50% of the follow-up period. Competitive employment is defined as a job receiving regular wages in a setting that is not set aside, sheltered, or enclaved, that is, the same job could be held by people without a mental illness or disability and is not a set-aside job in the TWP program. Secondary outcomes will include change in other occupational outcomes, PTSD symptoms, self esteem, community integration, and quality of life. We will explore the differences between groups in terms of occurrences of negative health outcomes.

These findings would provide generalizable evidence of the effectiveness of differing employment support to the VHA stakeholders who inform policy and service delivery for Veterans with PTSD. Given the number of Veterans with PTSD, it is of critical importance for the VA to offer employment service programs based on the best evidence-based recovery-oriented model for this group. Conducting a large multi-site study is the next logical step in confirming IPS as an evidence-based employment service for Veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Age greater than or equal to 18* (*18 or 19 depending on state legal definition of a minor) to age 65
* Eligible for VA TWP services
* Diagnosis of PTSD, as confirmed by Clinician Administered PTSD Scale (CAPS)
* Currently unemployed (and not participating in TWP - Impact Statement #3 10/4/13)
* Expression of interest in competitive employment (part-time or full-time - Impact Statement #3 10/4/13)
* Willing and able to give informed consent

Exclusion Criteria:

* Lifetime diagnosis if (i) schizophrenia, (ii) schizoaffective or (iii) bipolar I disorder
* Diagnosis of dementia or severe cognitive disorder (evidenced in the medical record)
* Unlikely that participant can complete the study; reasons may include: expected deployment, expected incarceration, expected long-term hospitalization, or expected relocation from the vicinity of the participating medical center (PMC) during the study period
* Active suicidal or homicidal ideation
* Current participation in another interventional trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2013-12-31 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2017-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Lynne Davis, MD AB, Study Chair — Tuscaloosa VA Medical Center, Tuscaloosa, AL
Locations (13):
- United States (13):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis LL, Resnick SG, Maieritsch KP, Weber KC, Erbes CR, Strom TQ, McCall KP, Kyriakides TC. Employment outcomes from VA vocational services involving transitional work for veterans with a diagnosis of posttraumatic stress disorder. Psychiatr Rehabil J. 2019 Sep;42(3):257-267. doi: 10.1037/prj0000357. Epub 2019 Apr 4. PMID 30945920
- [Derived] Mueller L, Wolfe WR, Neylan TC, McCaslin SE, Yehuda R, Flory JD, Kyriakides TC, Toscano R, Davis LL. Positive impact of IPS supported employment on PTSD-related occupational-psychosocial functional outcomes: Results from a VA randomized-controlled trial. Psychiatr Rehabil J. 2019 Sep;42(3):246-256. doi: 10.1037/prj0000345. Epub 2019 Apr 1. PMID 30932508
- [Derived] Davis LL, Kyriakides TC, Suris AM, Ottomanelli LA, Mueller L, Parker PE, Resnick SG, Toscano R, Scrymgeour AA, Drake RE; VA CSP #589 Veterans Individual Placement and Support Toward Advancing Recovery Investigators. Effect of Evidence-Based Supported Employment vs Transitional Work on Achieving Steady Work Among Veterans With Posttraumatic Stress Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Apr 1;75(4):316-324. doi: 10.1001/jamapsychiatry.2017.4472. PMID 29490371

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Individual Placement and Support (IPS): Individual Placement & Support: IPS uses an integrated "place-train" approach to help people obtain and maintain community-based competitive employment in their chosen occupation.
Period: Overall Study
Arm/Group | 1 Individual Placement and Support (IPS) | VA Transitional Work Program (TWP)
Started | 271 | 270
Completed | 250 (Primary Outcome Assessed over 18 months) | 240 (Primary Outcome assessed over 18 months)
Not Completed | 21 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Placement and Support (IPS) | VA Transitional Work Program (TWP) | Total
Number analyzed (Participants) | 271 | 270 | 541
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (10.7) | 41.9 (11.2) | 42.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 52 | 99
  Male | 224 | 218 | 442
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 43 | 47 | 90
  Not Hispanic or Latino | 228 | 223 | 451
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Responses to this question were collected from the participants. Some participants indicated more than one value; since this is a participant-reported variable, selecting one (primary) race/ethnicity indicator would not be appropriate.
  Participants
    White | 138 | 136 | 274
    African American | 115 | 110 | 225
    All Other | 32 | 36 | 68
    More than one race | 13 | 12 | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 271 | 270 | 541
Education Level [Count of Participants; unit: Participants]
  Less than High School | 1 | 4 | 5
  High School Diploma | 53 | 39 | 92
  Some College Credit | 106 | 118 | 224
  Associate's Degree | 55 | 35 | 90
  Bachelor's Degree | 40 | 57 | 97
  Master's or Doctoral Degree | 16 | 17 | 33
Housing Status [Count of Participants; unit: Participants]
  Single Family Home | 122 | 121 | 243
  Townhouse/Apartment/Condo | 91 | 94 | 185
  Other Housing | 16 | 20 | 36
  Inaquate Housing | 42 | 35 | 77
Inadequate Housing Status [Count of Participants; unit: Participants]
  Transitional Housing | 23 | 23 | 46
  Homeless Shelter or other | 19 | 12 | 31
Years of Homelessness [Mean (Standard Deviation); unit: Years] | 1.9 (1.7) | 1.9 (2.8) | 1.9 (2.0)
Time at Current Residence [Mean (Standard Deviation); unit: Years] — If housing was reported as adequate, this provides the time at that residence Population: The Time at Current Residence was reported for participants who indicated adequate housing
  Years
    number analyzed (Participants) | 229 | 235 | 464
    (all) | 3.6 (5.7) | 3.7 (6.2) | 3.6 (5.9)
Marital Status [Count of Participants; unit: Participants]
  Married | 89 | 84 | 173
  Divorced | 82 | 79 | 161
  Never Married | 68 | 67 | 135
  Separated/Cohabitating/widowed | 32 | 40 | 72
Length of current unemployment [Mean (Standard Deviation); unit: Years] | 2.7 (3.5) | 2.9 (4.1) | 2.8 (3.8)
Duration of longest job in lifetime [Mean (Standard Deviation); unit: years] | 8.3 (5.8) | 8.7 (6.4) | 8.5 (6.1)
Current Major Depressive Episode [Count of Participants; unit: Participants] | 87 | 83 | 170
Past Major Depressive Episode [Count of Participants; unit: Participants] | 183 | 173 | 356
Current Agoraphobia [Count of Participants; unit: Participants] | 64 | 59 | 123
Current Panic Disorder [Count of Participants; unit: Participants] | 37 | 33 | 70
Social Anxiety Disorder (generalized) [Count of Participants; unit: Participants] | 35 | 28 | 63
Alcohol Use disorder past 12 months [Count of Participants; unit: Participants] | 54 | 78 | 132
Non-alcohol use disorder past 12 months [Count of Participants; unit: Participants] — This measure includes Substance Dependence and Substance Abuse
  Participants | 47 | 40 | 87
Duration of PTSD [Mean (Standard Deviation); unit: years] | 13.3 (11.6) | 13.4 (11.3) | 13.3 (11.4)
Total CAPS-IV lifetime [Mean (Standard Deviation); unit: units on a scale] — Clinician Administered PTSD Scale (CAPS) Range: 0-136 (higher score is worse)
  units on a scale | 84.1 (18.9) | 84.8 (18.3) | 84.5 (18.6)
Current (last month) PTSD Checklist (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — Self-report PTSD Checklist for DSM-5 Range: 0 to 80 (higher score is worse)
  units on a scale | 46.2 (15.8) | 45.1 (17.0) | 45.6 (16.4)
PTSD Checklist (PCL-5) at current diagnostic threshold [Count of Participants; unit: Participants] — Number of participants with PTSD Checklist (PCL-5) score at or above the PTSD diagnostic threshold of 33
  Participants | 209 | 204 | 413
PCL-5 Current Severity [Count of Participants; unit: Participants] — Range: 0 to 80 (higher score is worse)
  Participants
    Very Mild (0-18) | 14 | 20 | 34
    Mild (19-37) | 64 | 60 | 124
    Moderate (38-59) | 128 | 138 | 266
    Severe (60-80) | 63 | 49 | 112

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Obtained and Maintained Competitive Employment for at Least 50% of the Active Follow-up Period
Description: The primary outcome will be achievement of a "steady worker" status, defined as obtaining and maintaining competitive employment for at least 50% of the active follow-up period (i.e., greater than or equal to 39 weeks).
Time Frame: 78 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Placement and Support (IPS) | VA Transitional Work Program (TWP)
Number analyzed (Participants) | 271 | 270
Participants | 105 | 63
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs VA Transitional Work Program (TWP); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.14, 95% CI 2-sided [1.46 to 3.14]

2. Secondary Outcome: Cumulative Gross Income
Description: Cumulative Gross Income is collected using the Employment Calendar source document and Employment Calendar Reconciliation case report form used for the primary outcome ascertainment. When possible, the CRC verifies income earned by reviewing paycheck stubs that the participant is instructed to maintain with the Employment Calendar.
Time Frame: Weekly for 78 weeks
Measure: Median (Inter-Quartile Range); unit: Dollars
Arm/Group | Individual Placement and Support (IPS) | VA Transitional Work Program (TWP)
Number analyzed (Participants) | 271 | 270
Dollars | 7290 [0 to 23174] | 1886 [0 to 17167]
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS) vs VA Transitional Work Program (TWP); Test type: Superiority; p = 0.004, Kruskal-Wallis; Site used as strata

3. Secondary Outcome: Change in PCL-5 Score of PTSD Symptoms
Description: PTSD Symptoms are assessed every three months during the follow-up period using the self-report PTSD Checklist (PCL-5) that the participant completes during the follow-up visits. Range of values 0-80 (higher score is worse).
Time Frame: 18-months (Change from baseline)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Individual Placement and Support (IPS) | VA Transitional Work Program (TWP)
Number analyzed (Participants) | 271 | 270
units on a scale | -3.66 [-6.09 to -1.23] | -0.82 [-3.24 to 1.59]
Statistical Analysis 1: Comparison: Individual Placement and Support (IPS); Test type: Other — Longitudinal analysis of PCL-5 (change from baseline); p = 0.07, Mixed Models Analysis; Mean Difference (Net) = -1.90, 95% CI 2-sided [-3.91 to 0.12]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a period of 18 months for each participant. Active monitoring of adverse events was initiated as soon as the study participant was randomized and continued to 30 days post-study follow-up.
Arm/Group | Individual Placement and Support (IPS) | VA Transitional Work Program (TWP)
All-Cause Mortality (participants affected / at risk) | 3/271 | 2/270
Serious Adverse Events (participants affected / at risk) | 63/271 | 64/270
Other Adverse Events (participants affected / at risk) | 36/271 | 40/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individual Placement and Support (IPS) (N=271) | VA Transitional Work Program (TWP) (N=270)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (2) | 0 (0)
Papilloedema (Eye disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 4 (5)
Death (General disorders) | 1 (1) | 0 (0)
Drug withdrawal syndrome (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (7) | 3 (3)
Chemical injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contrast media reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign intracranial hypertension (Nervous system disorders) | 1 (2) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiplegic migraine (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Postictal paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (2) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (2) | 1 (2)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Dependence (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Drug abuse (Psychiatric disorders) | 0 (0) | 3 (3)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 5 (9) | 3 (3)
Major depression (Psychiatric disorders) | 0 (0) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 2 (2) | 2 (2)
Psychotic behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Substance abuse (Psychiatric disorders) | 1 (1) | 2 (3)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 17 (29) | 17 (19)
Suicide attempt (Psychiatric disorders) | 4 (5) | 5 (6)
Priapism (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alcohol use (Social circumstances) | 1 (1) | 0 (0)
Physical assault (Social circumstances) | 0 (0) | 1 (1)
Victim of crime (Social circumstances) | 0 (0) | 1 (1)
Victim of homicide (Social circumstances) | 0 (0) | 1 (1)
Alcohol detoxification (Surgical and medical procedures) | 3 (6) | 0 (0)
Detoxification (Surgical and medical procedures) | 0 (0) | 1 (1)
Drug detoxification (Surgical and medical procedures) | 1 (1) | 0 (0)
Elective surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 1 (1)
Self-medication (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (4)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individual Placement and Support (IPS) (N=271) | VA Transitional Work Program (TWP) (N=270)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Chemical eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to violent event (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Aggression (Psychiatric disorders) | 2 (2) | 2 (2)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (5) | 1 (2)
Dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Flashback (Psychiatric disorders) | 2 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 2 (2) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (2) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 3 (3) | 3 (3)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Self-injurious ideation (Psychiatric disorders) | 0 (0) | 0 (0)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 11 (13) | 5 (7)
Violence-related symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hair disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alcohol use (Social circumstances) | 1 (1) | 0 (0)
Loss of employment (Social circumstances) | 0 (0) | 1 (1)
Stress at work (Social circumstances) | 0 (0) | 1 (1)
Verbal abuse (Social circumstances) | 0 (0) | 1 (1)
Victim of abuse (Social circumstances) | 0 (0) | 1 (2)
Victim of sexual abuse (Social circumstances) | 1 (1) | 1 (1)
Alcohol detoxification (Surgical and medical procedures) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes